CLINICAL TRIAL: NCT04535531
Title: A Phase 3 Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study Comparing the Efficacy and Safety of SB206 and Vehicle Gel Once Daily in the Treatment of Molluscum Contagiosum
Brief Title: A Phase 3 Molluscum Contagiosum Efficacy and Safety Study
Acronym: B-SIMPLE4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novan, Inc. (Industry)
Collaborators: Therapeutics, Inc. (Industry); Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NI-MC304
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-11

CONDITIONS: Molluscum Contagiosum
MeSH Terms: conditions — Molluscum Contagiosum | interventions — berdazimer sodium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SB206 10.3% berdazimer (Experimental): SB206 10.3% berdazimer topically once daily
  Interventions: Drug: SB206 10.3% berdazimer
- vehicle gel (Placebo Comparator): Vehicle gel topically once daily
  Interventions: Drug: vehicle gel

INTERVENTIONS:
Drug: SB206 10.3% berdazimer — Topically once daily
  Other Names: SB206 12% berdazimer sodium
  Arms: SB206 10.3% berdazimer
Drug: vehicle gel — Topically once daily
  Arms: vehicle gel

SUMMARY:
This is a phase 3 multi-center, randomized, double-blind, vehicle-controlled, parallel group study to be conducted in up to approximately 850 subjects 6 months of age and older with molluscum contagiosum (MC). Subjects or their caregivers will apply SB206 10.3% or Vehicle Gel once daily for a minimum of 4 weeks and up to 12 weeks to all lesions identified at Baseline and new treatable lesions that arise during the course of the study.

DETAILED DESCRIPTION:
This is a phase 3 multi-center, randomized, double-blind, vehicle-controlled, parallel group study to be conducted in up to approximately 850 subjects 6 months of age and older with molluscum contagiosum (MC). After obtaining informed consent/assent, subjects who satisfy entry criteria will be randomized 1:1 (active:vehicle). Subjects receiving current treatment for MC at the time of the Screening Visit will enter a wash out period of up to 14 days prior to randomization.

Subjects or their caregivers will apply treatment once daily to all lesions identified at Baseline and new lesions that arise during treatment for a minimum of 4 weeks and up to 12 weeks. If the investigator determines all lesions are cleared at a visit, the treatment may stop. If treatment is stopped due to clearance, subjects will continue regularly scheduled visits through Week 24/ET2. Study drug will be dispensed through Week 12/ET1 in case of lesion recurrence between study visits. At each visit subsequent to stopping treatment due to clearance, the investigator will determine if new lesions have occurred since the last visit, and if so, the subject or caregiver will be instructed by the investigator to re-initiate treatment. If the subject or caregiver see new lesions or re-occurrence of lesions in between visits, they should treat these lesions until the next visit. No study drug will be provided after the Week 12 visit. The subject or caregiver will apply study drug to the individual lesions. Periocular lesions will be treated if the lesions are at least 2 cm from the edge of the eye. Subjects will visit the clinic in person at Screening/Baseline, Week 2, Week 4 (unless visit is performed remotely), Week 8, Week 12, and Week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Be 6 months of age or older, and in good general health;
2. Have a documented informed consent form signed by subject or a parent or legal guardian and an assent form as required;
3. Have between 3 and 70 treatable MC lesions at Baseline;
4. For women of childbearing potential (WOCBP): Must have a negative urine pregnancy test prior to randomization and must agree to use an effective method of birth control during the study; Note: WOCBP and effective methods of birth control are outlined in Section 9.4.
5. Have a device (phone, tablet, personal computer, etc.) that will support remote visits, including a camera;
6. Be willing and able to follow study instructions and likely to complete all study requirements, including remote study visits.

Exclusion Criteria:

1. Have strongly suggested sexually transmitted MC and do not agree to refrain from sexual activities throughout the study period;
2. Are immunosuppressed, have immunodeficiency disorder, or are on immunosuppressive treatment;
3. Have significant injury on and/or surrounding MC that may impact ability to treat and count lesions;
4. Have received treatment with topical calcineurin inhibitors or steroids on MC or within 2 cm of MC lesions within 14 days prior to Baseline;
5. Have received treatment for MC during the 14 days prior to Baseline with podophyllotoxin, imiquimod, cantharidin, sinecatechins, topical retinoids, oral or topical zinc, or other homeopathic or over the counter (OTC) products including, but not limited to, ZymaDerm and tea tree oil, cimetidine and other histamine H2 receptor antagonists (including Zantac), or any agent that in the opinion of the investigator may be relevant - (e.g. wart therapies);
6. Have received surgical procedures related to MC (e.g. cryotherapy, curettage) within 14 days prior to Baseline;
7. Have MC only in periocular area;
8. Female subjects who are pregnant, planning a pregnancy or breastfeeding;
9. Have known hypersensitivity to any ingredients of SB206 or Vehicle Gel including excipients;
10. Have participated in a previous study with a berdazimer containing product (i.e. SB204, SB206, SB208, SB414);
11. Have more than one other family member participating in this study (NI-MC304);
12. Have at least 1 family member currently participating in a study, other than this study, with a berdazimer containing product (i.e. SB204, SB206, SB208, SB414);
13. Have participated in any other trial of an interventional investigational drug or device within 14 days or concurrent participation in another interventional research study;
14. History or presence of clinically significant medical, psychiatric, or emotional condition that, in opinion of the investigator, would compromise the safety of the subject or the quality of the data.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 891 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Maeda Chubachi, MD PhD, Study Director — Novan, Inc.
Locations (55):
- United States (55):
  - Site #312, Glendale, Arizona
  - Site #101, Hot Springs, Arkansas
  - Site #272, Rogers, Arkansas
  - Site #336, Fountain Valley, California
  - Site #329, Fremont, California
  - Site# 348, Fresno, California
  - Site #161, San Diego, California
  - Site #327, Thousand Oaks, California
  - Site #325, Greenwood Village, Colorado
  - Site #335, Apopka, Florida
  - Site #342, Boca Raton, Florida
  - Site #333, Fort Lauderdale, Florida
  - Site #334, Homestead, Florida
  - Site #278, Miami, Florida
  - Site #314, Miami Lakes, Florida
  - Site #341, Orlando, Florida
  - Site #227, Sanford, Florida
  - Site #305, Tampa, Florida
  - Site #116, Newnan, Georgia
  - Site #340, Chicago, Illinois
  - Site #253, Rolling Meadows, Illinois
  - Site #288, Evansville, Indiana
  - Site #310, Plainfield, Indiana
  - Site #328, Bowling Green, Kentucky
  - Site #347, Lexington, Kentucky
  - Site # 117, Louisville, Kentucky
  - Site #294, Owensboro, Kentucky
  - Site #321, Baton Rouge, Louisiana
  - Site# 349, Covington, Louisiana
  - Site #332, New Orleans, Louisiana
  - Site #297, New Orleans, Louisiana
  - Site #330, Rockville, Maryland
  - Site #346, Brighton, Massachusetts
  - Site #274, Clarkston, Michigan
  - Site #121, New Brighton, Minnesota
  - Site #338, Omaha, Nebraska
  - Site #201, Berlin, New Jersey
  - Site #331, Verona, New Jersey
  - Site #279, Greensboro, North Carolina
  - Site #250, Portland, Oregon
  - Site #265, Sugarloaf, Pennsylvania
  - Site #311, Warwick, Rhode Island
  - Site #295, Fountain Inn, South Carolina
  - Site #255, Summerville, South Carolina
  - Site #291, Kingsport, Tennessee
  - Site #326, Knoxville, Tennessee
  - Site #316, Murfreesboro, Tennessee
  - Site #337, Houston, Texas
  - Site #299, Longview, Texas
  - Site #224, San Antonio, Texas
  - Site #281, Layton, Utah
  - Site #345, West Jordan, Utah
  - Site #267, Richmond, Virginia
  - Site #339, Spokane, Washington
  - Site #343, Morgantown, West Virginia

REFERENCES:
- [Derived] Browning JC, Cartwright M, Thorla I Jr, Martin SA, Olayinka-Amao O, Maeda-Chubachi T. A Patient-Centered Perspective of Molluscum Contagiosum as Reported by B-SIMPLE4 Clinical Trial Patients and Caregivers: Global Impression of Change and Exit Interview Substudy Results. Am J Clin Dermatol. 2023 Jan;24(1):119-133. doi: 10.1007/s40257-022-00733-9. Epub 2022 Oct 26. PMID 36287306
- [Derived] Browning JC, Enloe C, Cartwright M, Hebert A, Paller AS, Hebert D, Kowalewski EK, Maeda-Chubachi T. Efficacy and Safety of Topical Nitric Oxide-Releasing Berdazimer Gel in Patients With Molluscum Contagiosum: A Phase 3 Randomized Clinical Trial. JAMA Dermatol. 2022 Aug 1;158(8):871-878. doi: 10.1001/jamadermatol.2022.2721. PMID 35830173

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects receiving current treatment for MC at the time of the Screening Visit entered a wash out period of up to 14 days prior to randomization.
Period: Overall Study
Arm/Group | SB206 10.3% Berdazimer | Vehicle Gel
Started | 444 | 447
Completed | 363 | 390
Not Completed | 81 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB206 10.3% Berdazimer | Vehicle Gel | Total
Number analyzed (Participants) | 444 | 447 | 891
Age, Customized [Number; unit: participants]
  <1 year old | 1 | 0 | 891
  1 to <2 years old | 15 | 12 | 27
  2 years old to <6 years old | 220 | 213 | 433
  6 years old to <12 years old | 178 | 201 | 379
  12 years old to <18 years old | 24 | 15 | 39
  18 years old | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 234 | 450
  Male | 228 | 213 | 441
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 94 | 87 | 181
  Not Hispanic or Latino | 345 | 357 | 702
  Ethnicity Not Reported | 4 | 1 | 5
  Unknown | 1 | 2 | 3
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 6 | 6 | 12
  Black or African American | 21 | 28 | 49
  Native Hawaiian or Other Pacific Islander | 4 | 2 | 6
  White | 387 | 382 | 769
  More than One Race | 13 | 13 | 26
  Race Not Reported | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  United States | 444 | 447 | 891
Baseline number of Molluscum lesions [Mean (Standard Deviation); unit: Molluscum lesions] | 23.1 (17.60) | 20.5 (16.18) | 21.8 (16.94)

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance of All Treatable MC at Week 12
Description: Percent (proportion) of subjects with complete clearance of all treatable MC at Week 12. This was measured by dividing the number of subjects who showed complete clearance by the number in that treatment group (this represents our primary outcome variable).
Time Frame: 12 Weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Groups:
- SB206: SB206 gel applied topically, once daily for 12 weeks.
- Placebo: Placebo gel applied topically, once daily for 12 weeks.
Arm/Group | SB206 | Placebo
Number analyzed (Participants) | 444 | 447
Participants | 144 | 88

2. Secondary Outcome: A Lesion Count of 0 or 1 of All Treatable MC at Week 12
Description: Percent (proportion) of subjects achieving a lesion count of 0 or 1 of all treatable MC at Week 12.
Time Frame: 12 Weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | SB206 | Placebo
Number analyzed (Participants) | 444 | 447
Participants | 193 | 110

3. Secondary Outcome: 90% Reduction From Baseline in the Number of All Treatable MC at Week 12
Description: Percent (proportion) of subjects achieving at least a 90% reduction from Baseline in the number of all treatable MC at Week 12
Time Frame: 12 Weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | SB206 | Placebo
Number analyzed (Participants) | 444 | 447
Participants | 191 | 107

4. Secondary Outcome: Complete Clearance of All Treatable MC at Week 8
Description: Percent (proportion) of subjects with complete clearance of all treatable MC at Week 8. This was measured by dividing the number of subjects who showed complete clearance at week 8 by the number in that treatment group (this represents our secondary outcome variable).
Time Frame: 8 Weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | SB206 | Placebo
Number analyzed (Participants) | 444 | 447
Participants | 87 | 52

5. Secondary Outcome: Change From Baseline in the Number of All Treatable MC at Week 4
Description: Percent change from Baseline in the number of all treatable MC at Week 4
Time Frame: 4 Weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | SB206 | Placebo
Number analyzed (Participants) | 444 | 447
percentage of change from baseline | -25.5 (2.86) | -9.2 (2.86)

ADVERSE EVENTS:
Time Frame: Baseline visit to end of study visit, 84 days.
Description: Only TEAE were to be considered.
Arm/Group | SB206 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/444 | 0/447
Serious Adverse Events (participants affected / at risk) | 0/444 | 1/447
Other Adverse Events (participants affected / at risk) | 221/444 | 37/447
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB206 (N=444) | Placebo (N=447)
Supracondylar Fracture of right humerus, closed reduction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Moderate/unrelated/hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB206 (N=444) | Placebo (N=447)
Application site pain (General disorders) | 83 (113) | 23 (26)
Application site erythema (General disorders) | 52 (66) | 6 (7)
Application site pruritus (General disorders) | 33 (38) | 5 (5)
Application site exfoliation (General disorders) | 27 (45) | 0 (0)
Application site dermatitis (General disorders) | 26 (28) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must wait 18 months after the closeout of the trial at all Study sites or until the publication of the multi-site Sponsor results. The only restriction on PI publication after that time is that the sponsor can review results communications prior to public release and can request confidential or proprietary information be removed or can embargo communications regarding trial results for a period that is more than 90 days but less than 120 days.

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT04535531/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/31/NCT04535531/SAP_001.pdf